CLINICAL TRIAL: NCT03343106
Title: Combining Acceptance and Commitment Therapy With Exposure and Response Prevention to Enhance Treatment Engagement in Obsessive-Compulsive Disorder
Brief Title: Combining Acceptance and Commitment Therapy With Exposure and Response Prevention to Enhance Treatment Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); International OCD Foundation (Unknown)
Responsible Party: Principal Investigator, Michael Twohig, Ph.D., Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2965
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Acceptance and Commitment Therapy; Exposure and Response Prevention; Psychotherapy; Obsessive-Compulsive Disorder; Treatment Acceptability; Treatment Adherence
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT plus ERP (Experimental): Sessions 1 and 2 involved information-gathering, discussion of the ACT model of OCD and ERP, and introduction to self-monitoring of rituals. Session 3 involved the development of an exposure hierarchy and response prevention plan, and further explanation of the ACT-based approach to ERP which focuses on learning flexible responding in the presence of obsessions, anxiety, and urges to ritualize. Exposure practices (sessions 4-16) were procedurally similar to the ERP condition, but focused on the facilitation of ACT processes rather than on fear extinction. Homework exposure practice was linked to the participant's goals and values. Session 16 included an ACT model of relapse prevention focusing on following one's values in the presence of obsessive thoughts and compulsive urges.
  Interventions: Behavioral: ACT plus ERP
- ERP alone (Experimental): ERP followed Kozak and Foa's treatment manual. Sessions 1 and 2 included information-gathering, psychoeducation about the cognitive-behavioral model of OCD and rationale for ERP, and introduction to self-monitoring of rituals. Session 3 was dedicated to developing the treatment plan (exposure hierarchy, response prevention plan). Sessions 4-16 included in-session prolonged and repeated gradual exposure therapy (in vivo and imaginal as needed), the assignment of daily exposure practices for between-sessions, and instructions to refrain from rituals (response prevention in session and between sessions), along with self monitoring of any rituals that were performed. Session 16 also addressed discontinuation and relapse prevention.
  Interventions: Behavioral: ERP alone

INTERVENTIONS:
Behavioral: ACT plus ERP — 16 twice-weekly sessions of 120-minute individual psychotherapy consisting of Acceptance and Commitment Therapy plus Exposure and Response Prevention (ACT plus ERP).
  Arms: ACT plus ERP
Behavioral: ERP alone — 16 twice-weekly sessions of 120-minute individual psychotherapy consisting of Exposure and Response Prevention (ERP alone) monotherapy.
  Arms: ERP alone

SUMMARY:
The aim of the study was to evaluate whether integrating Acceptance and Commitment Therapy (ACT) with Exposure and Response Prevention (ERP) increases the acceptability, tolerability, and adherence with ERP techniques relative to ERP without ACT. Fifty-eight adults with a DSM-IV diagnosis of Obsessive-Compulsive Disorder (OCD) received 16 twice-weekly sessions (2 hours per session) of either ERP with the inclusion of ACT techniques (ERP+ACT; n = 30) or ERP alone (n = 28). Assessments using interviews, self-report questionnaires, and behavioral observations were conducted at pre- and post-test, and at 6 month follow-up. Specific hypotheses were: 1) Patients receiving ERP+ACT will report greater treatment acceptability, and show higher quantity and quality of completed self-directed ERP assignments, relative to patients receiving standard ERP; 2) Both ERP and ERP+ACT will lead to clinically significant reductions in OCD symptoms from pre- to post-test and from pre-test to follow-up.

DETAILED DESCRIPTION:
1. BACKGROUND AND SIGNIFICANCE.

   The most effective psychological treatment for Obsessive-Compulsive Disorder (OCD) is Exposure and Response Prevention (ERP), which entails confronting obsessional triggers (i.e., exposure) and resisting urges to ritualize (response prevention). Although successful, these techniques are challenging and provoke high levels of anxiety. This may contribute to the fact that between 25% and 50% of patients with access to ERP refuse treatment, drop out prematurely, or do not adhere to the treatment instructions and show attenuated response. Given the effectiveness of ERP techniques, developing ways to make them more tolerable and increase patient adherence, while not compromising therapeutic integrity, is an important next step in OCD treatment research. Recent investigations have addressed whether adding medications, cognitive therapy, or motivational Interviewing to ERP improves outcome and adherence; yet to date, no consensus has emerged regarding the degree to which these combination treatments are more effective than ERP monotherapy. Acceptance and Commitment Therapy (ACT), which has recently been studied for OCD, offers new hope for addressing the tolerability and adherence issues with ERP. Specifically, ACT uses acceptance and mindfulness processes to foster a willingness to experience unwanted inner experiences (e.g., obsessional thoughts, anxiety). These acceptance and mindfulness processes are consistent with ERP, but they are hypothesized to increase engagement in exposure exercises beyond ERP alone. There is evidence for this claim from a randomized trial which demonstrated that ACT, without in-session exposure, had clinical response rates in the 55-65% range at posttreatment and three month follow-up using an intent to treat analysis. Additionally, drop-out and refusal rates were low at 12.2% and treatment acceptability at posttreatment was near the maximum on the scale 4.3 out of 5. In this study, for experimental reasons, ACT did not include in-session ERP. However, the most theoretically and practically consistent use of ACT for OCD is as a context from which to conduct exposure therapy or ERP. While ACT focuses on processes (e.g., acceptance, defusion, values) that are distinct from those involved in ERP (e.g., habituation, cognitive change), an important goal of both treatments is to broaden the patient's engagement with feared stimuli. In fact, ACT procedures have been shown to increase involvement in difficult activities, including participating in exposure therapy for anxiety disorders and willingness to experience unwanted obsessive thoughts. Thus, building ACT techniques into ERP is likely to help patients (a) engage in ERP tasks, (b) confront high levels of anxiety without using escape/avoidance strategies, and (c) resist rituals. The aim of the proposed study is to evaluate whether integrating ACT increases the acceptability, tolerability, and adherence with ERP techniques relative to ERP without ACT.
2. STUDY DESIGN AND HYPOTHESES.

   Fifty-eight adults with a DSM-IV diagnosis of Obsessive-Compulsive Disorder (OCD) received 16 twice-weekly sessions (2 hours per session) of either ERP with the inclusion of ACT techniques (ERP+ACT; n = 30) or ERP alone (n = 28). Assessments using interviews, self-report questionnaires, and behavioral observations were conducted at pre- and post-test, and at 6 month follow-up. Specific hypotheses were: 1) Patients receiving ERP+ACT will report greater treatment acceptability, and show higher quantity and quality of completed self-directed ERP assignments, relative to patients receiving standard ERP; 2) Both ERP and ERP+ACT will lead to clinically significant reductions in OCD symptoms from pre- to post-test and from pre-test to follow-up.
3. METHODS

3a. Sample Size and Recruitment. The investigators aimed for an intent-to-treat sample of 60 adults across two sites: The Center for Clinical Research at Utah State University (USU) and the Anxiety and Stress Disorders Clinic at the University of North Carolina, Chapel Hill (UNC). Patients were recruited via advertisement of the study and via referrals from primary care and mental health providers familiar with the treatment centers. The USU Center (Twohig) and the UNC Clinic (Abramowitz) are well known research-oriented treatment clinics in their regions. USU is within a 1:30 minute drive of two million people and travel for treatment is common given the rural nature of the area. Also, no other known entity recruits participants with OCD in this area. The Raleigh-Durham-Chapel Hill area of NC is home to over one million people, and the UNC Clinic receives a steady stream of inquiries for treatment. Patient advocacy groups and associations that post research trials on the Internet were contacted to further publicize the study.

3b. Establishing Diagnoses. All diagnoses were established by trained interviewers using the Mini International Neuropsychiatric Interview (MINI).

3c. Randomization to Treatment Groups. Subsequent to screening, 30 individuals were randomly assigned (using a random number generator) to receive ERP+ACT and 28 to receive ERP monotherapy. With the exception of the inclusion of ACT techniques in the ERP+ACT condition, treatment was identical across the two groups (i.e., the number and duration of exposure sessions were the same).

3d. Treatments. ERP. ERP treatment was manualized based on Kozak and Foa's protocol and included 16 twice-weekly 120 minute sessions. Therapists were advanced graduate students who had received extensive training from experts in ERP and ACT for OCD. Sessions 1 and 2 included information-gathering, psychoeducation, presentation of the rationale for ERP, and introduction to self-monitoring of rituals. Session 3 was dedicated to developing the treatment plan (exposure hierarchy, response prevention plan). Sessions 4-15 included in-session prolonged and repeated gradual exposure therapy, informal discussion of mistaken cognitions, daily exposure homework assignments, and instructions to refrain from rituals (response prevention in session and between sessions), along with self monitoring of any rituals that were performed. Session 16 addressed discontinuation and relapse prevention.

ACT+ERP. This condition matched the ERP condition in terms of the number and duration of exposure sessions. Sessions 1 and 2 involved an abbreviated discussion of the ACT model of ERP focusing on acceptance of obsessions and anxiety, just noticing and not acting on obsessions, being present with one's internal experiences, and linking therapy to one's values. Session 3 involved the development of an exposure hierarchy and response prevention plan, and explaining the ACT-based approach to ERP which focuses on learning flexible responding in the presence of obsessions, anxiety, and urges to ritualize. The exposure exercises were procedurally similar to ERP but focused on the facilitation of ACT processes. For example, the therapist might teach just noticing of obsessions by exposing the participant to the feared stimulus and asking the participant to watch the obsessional thoughts pass by as if they were leaves floating on a stream. Homework exposure practice was linked to the patient's goals and values, and participants were instructed to practice ACT processes during these assignments. Session 16 covered an ACT-based model of relapse prevention focusing on following one's values in the presence of obsessive thoughts and compulsive urges.

3e. Standardization and Integrity Procedures. All assessors and therapists were trained to competency in their duties by Drs. Twohig and Abramowitz. All assessment and treatment sessions were videotaped and a random selection of 20% of tapes were reviewed by the investigators and scored for integrity of implementation. Drs. Twohig and Abramowitz also served as supervisors on the project. Cross-site data and video sharing of supervision occurred via the Internet in a HIPAA-compliant manner and weekly meetings occurred via Skype.

3f. Length of Study. The length of the study was 6 years. The investigators developed the ERP+ACT treatment manual during the first two months of the study period. Following this, the investigators completed recruitment and treatment of all patients between the 1st and 6th years. This left the final 1 year for follow-up data collection, data analysis, and for writing up and presenting the results.

3g. Statistical Methods. The investigators will use the following procedures to address each hypotheses: 1) Between-groups t-tests to examine differences on measures of treatment acceptability and the quantity and quality of adherence to ERP assignments at post-treatment. Corresponding effect sizes will be computed to examine the magnitude of this effect. 2) Within-group t-tests to determine the statistical significance of pre-posttest and pretest-follow-up differences on outcome measures. Corresponding within-group effect sizes will also be computed to examine the magnitude of these differences. Further, the methods described by Jacobson & Truax to examine the extent of clinically significant and reliable change from pre to posttest and at follow-up will be utilized.

3h. Power Analyses. Power calculations were based on the average within-group effect size of 1.41 reported in a meta-analysis of CBT for OCD. This effect size was derived from clinical interview measures (e.g., the Yale-Brown Obsessive Compulsive Scale). A sample size of 60 affords greater than 90% power to detect a similar effect size with a t-test in the present study if alpha is set at .05. There are no available studies comparing treatment adherence and quality of life between two active psychological treatments for OCD from which to calculate power estimates. The investigators will therefore examine effect sizes in addition to significance levels when comparing between ERP+ACT and ERP on these variables.

4. INTENDED USE OF THE RESULTS

The results from the present study will be published and disseminated through conference presentations. They will also be used as pilot data to apply for NIMH funding for a larger study using the R34 mechanism (treatment development).

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV-TR principal diagnosis of OCD for at least 1 year
* Willing to attend all 16 therapy sessions
* Fluent in English
* No previous Cognitive Behavior Therapy or Acceptance and Commitment Therapy for OCD
* If on medication for OCD, willing to remain at a fixed dose while participating in the study

Exclusion Criteria:

* Current severe depression or suicidal ideation
* Current substance abuse or dependence
* Current mania, psychosis, or borderline or schizotypal personality disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-07-12 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at 8 weeks | Posttreatment (8 weeks after Baseline)
  Global OCD severity was measured using the Y-BOCS, a semi-structured interview that includes a symptom checklist and 10-item severity scale. The checklist is first used to identify the patient's particular obsessions and compulsions. The severity scale then assesses the main obsessions (items 1-5) and compulsions (items 6-10) on the following five parameters: (a) time, (b) interference, (c) distress, (d) resistance, and (e) degree of control. The clinician rates each item from 0 (no symptoms) to 4 (extreme) based on the past week. The 10 items are added to produce a total severity score that ranges from 0 to 40. The Y-BOCS is the most widely used measure of OCD severity and has satisfactory psychometric properties. The internal consistency (Cronbach's alpha) of the pre-treatment Y-BOCS in the present sample was .74.
Change from Posttreatment Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at 6 months | Follow-up (6 months after the end of treatment)
  Global OCD severity was measured using the Y-BOCS, a semi-structured interview that includes a symptom checklist and 10-item severity scale. The checklist is first used to identify the patient's particular obsessions and compulsions. The severity scale then assesses the main obsessions (items 1-5) and compulsions (items 6-10) on the following five parameters: (a) time, (b) interference, (c) distress, (d) resistance, and (e) degree of control. The clinician rates each item from 0 (no symptoms) to 4 (extreme) based on the past week. The 10 items are added to produce a total severity score that ranges from 0 to 40. The Y-BOCS is the most widely used measure of OCD severity and has satisfactory psychometric properties. The internal consistency (Cronbach's alpha) of the pre-treatment Y-BOCS in the present sample was .74.

SECONDARY OUTCOMES:
Change from Baseline Beck Depression Inventory II (BDI-II) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The BDI-II is a 21-item self-report scale that assesses the severity of affective, cognitive, motivational, vegetative, and psychomotor components of depression. Scores of 10 or less are considered normal; scores of 20 or greater suggest the presence of clinical depression. The BDI has excellent reliability and validity and is widely used in clinical research. In the present sample, the pre-treatment BDI had a Cronbach's alpha of .93.
Change from Posttreatment Beck Depression Inventory II (BDI-II) at 6 months | Follow-up (6 months after the end of treatment)
  The BDI is a 21-item self-report scale that assesses the severity of affective, cognitive, motivational, vegetative, and psychomotor components of depression. Scores of 10 or less are considered normal; scores of 20 or greater suggest the presence of clinical depression. The BDI has excellent reliability and validity and is widely used in clinical research. In the present sample, the pre-treatment BDI had a Cronbach's alpha of .93.
Change from Baseline Acceptance and Action Questionnaire - II (AAQ-II) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The AAQ-II is a 7-item 7-point Likert-type measure of experiential avoidance/psychological inflexibility. The items reflect: (a) unwillingness to experience unwanted emotions and thoughts, and (b) the inability to be in the present moment and behave according to value-directed actions when experiencing unwanted psychological events. The AAQ-II shows good psychometric properties (mean alpha of .88). In present sample, the pre-treatment AAQ-II had a Cronbach's alpha of .87.
Change from Posttreatment Acceptance and Action Questionnaire - II (AAQ-II) at 6 months | Follow-up (6 months after the end of treatment)
  The AAQ-II is a 7-item 7-point Likert-type measure of experiential avoidance/psychological inflexibility. The items reflect: (a) unwillingness to experience unwanted emotions and thoughts, and (b) the inability to be in the present moment and behave according to value-directed actions when experiencing unwanted psychological events. The AAQ-II shows good psychometric properties (mean alpha of .88). In present sample, the pre-treatment AAQ-II had a Cronbach's alpha of .87.
Session-level Change in Acceptance and Action Questionnaire - II (AAQ-II) at each session | Sessions 1-16 (Twice per week for 8 weeks following Baseline)
  The AAQ-II is a 7-item 7-point Likert-type measure of experiential avoidance/psychological inflexibility. The items reflect: (a) unwillingness to experience unwanted emotions and thoughts, and (b) the inability to be in the present moment and behave according to value-directed actions when experiencing unwanted psychological events. The AAQ-II shows good psychometric properties (mean alpha of .88). In present sample, the pre-treatment AAQ-II had a Cronbach's alpha of .87.
Change from Baseline Distress Tolerance Scale (DTS) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The DTS is composed of 14 items answered on 5-point Likert-type scales ranging from 1, strongly agree, to 5, strongly disagree, evaluating participants' ability to experience and endure negative emotional states. Greater scores reflect higher levels of distress tolerance. This scale has good psychometric properties, including high internal consistency (α=.89) and appropriate convergence with other self-report ratings of affective distress and regulation. In addition, the DTS has demonstrated adequate 6-month test-retest reliability (r=.61). In the present sample, the pre-treatment DTS had a Cronbach's alpha of .94.
Change from Posttreatment Distress Tolerance Scale (DTS) at 6 months | Follow-up (6 months after the end of treatment)
  The DTS is composed of 14 items answered on 5-point Likert-type scales ranging from 1, strongly agree, to 5, strongly disagree, evaluating participants' ability to experience and endure negative emotional states. Greater scores reflect higher levels of distress tolerance. This scale has good psychometric properties, including high internal consistency (α=.89) and appropriate convergence with other self-report ratings of affective distress and regulation. In addition, the DTS has demonstrated adequate 6-month test-retest reliability (r=.61). In the present sample, the pre-treatment DTS had a Cronbach's alpha of .94.
Change from Baseline Interpretation of Intrusions Inventory (III) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The III is a semi-idiographic measure designed to assess negative appraisals of intrusive thoughts. The respondent reads a set of instructions that includes examples of intrusive thoughts (e.g., images of the baby lying dead in his crib, an impulse to shake the infant very hard) and then is asked to identify one or two examples of his or her own intrusions. The respondent then identifies the extent of his or her agreement with 31 items concerning various negative appraisals of these intrusions (e.g., "I would be a better person if I didn't have this thought"). Although 3 theoretically derived subscales were initially proposed: (a) importance of thoughts, (b) control of thoughts, and (c) responsibility, data suggests that only a single factor exists. The internal consistency of the pre-treatment III in the present sample was .94.
Change from Posttreatment Interpretation of Intrusions Inventory (III) at 6 months | Follow-up (6 months after the end of treatment)
  The III is a semi-idiographic measure designed to assess negative appraisals of intrusive thoughts. The respondent reads a set of instructions that includes examples of intrusive thoughts (e.g., images of the baby lying dead in his crib, an impulse to shake the infant very hard) and then is asked to identify one or two examples of his or her own intrusions. The respondent then identifies the extent of his or her agreement with 31 items concerning various negative appraisals of these intrusions (e.g., "I would be a better person if I didn't have this thought"). Although 3 theoretically derived subscales were initially proposed: (a) importance of thoughts, (b) control of thoughts, and (c) responsibility, data suggests that only a single factor exists. The internal consistency of the pre-treatment III in the present sample was .94.
Session-level Change in Interpretation of Intrusions Inventory (III) at each session | Sessions 1-16 (twice per week for 8 weeks following Baseline)
  The III is a semi-idiographic measure designed to assess negative appraisals of intrusive thoughts. The respondent reads a set of instructions that includes examples of intrusive thoughts (e.g., images of the baby lying dead in his crib, an impulse to shake the infant very hard) and then is asked to identify one or two examples of his or her own intrusions. The respondent then identifies the extent of his or her agreement with 31 items concerning various negative appraisals of these intrusions (e.g., "I would be a better person if I didn't have this thought"). Although 3 theoretically derived subscales were initially proposed: (a) importance of thoughts, (b) control of thoughts, and (c) responsibility, data suggests that only a single factor exists. The internal consistency of the pre-treatment III in the present sample was .94.
Change from Baseline Believability of Anxious Feelings and Thoughts Questionnaire (BAFT) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The BAFT is a self-report measure of cognitive fusion with anxious thoughts and feelings. It consists of 16 items representing different thoughts which are rated on a 7-point Likert-type scale ranging from 1 (not at all believable) to 7 (completely believable) to the extent that the individual believes in them. A hierarchical factor structure of the BAFT with three lower order factors and one hierarchical factor was found. The three lower order factors were labeled Somatic Concerns (fusion with somatic concerns), Emotion Regulation (fusion with excessive struggle with and control of emotions), and Negative Evaluation (fusion with negative evaluation of anxious thoughts and feelings). The internal consistency of the total pre-treatment BAFT in the present sample was .86. Individual subscale internal consistencies ranged from .72 to .77.
Change from Posttreatment Believability of Anxious Feelings and Thoughts Questionnaire (BAFT) at 6 months | Follow-up (6 months after the end of treatment)
  The BAFT is a self-report measure of cognitive fusion with anxious thoughts and feelings. It consists of 16 items representing different thoughts which are rated on a 7-point Likert-type scale ranging from 1 (not at all believable) to 7 (completely believable) to the extent that the individual believes in them. A hierarchical factor structure of the BAFT with three lower order factors and one hierarchical factor was found. The three lower order factors were labeled Somatic Concerns (fusion with somatic concerns), Emotion Regulation (fusion with excessive struggle with and control of emotions), and Negative Evaluation (fusion with negative evaluation of anxious thoughts and feelings). The internal consistency of the total pre-treatment BAFT in the present sample was .86. Individual subscale internal consistencies ranged from .72 to .77.
Change from Baseline Obsessive Beliefs Questionnaire (OBQ) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The OBQ is a 44-item self-report questionnaire developed to assess a variety of dysfunctional beliefs thought to underlie OCD symptoms. Three factor analytically derived subscales correspond to the following domains of obsessive beliefs: (a) overestimates of threat and responsibility for harm, (b) importance and control of intrusive thoughts, and (c) perfectionism and the need for certainty. Participants rate their agreement with each of 44 statements from 1 (disagree very much) to 7 (agree very much). The instrument possesses good validity and internal consistency, and has been widely studied in clinical and nonclinical samples. Cronbach alphas for the subscales ranged from .89 to .91.
Change from Posttreatment Obsessive Beliefs Questionnaire (OBQ) at 6 months | Follow-up (6 months after the end of treatment)
  The OBQ is a 44-item self-report questionnaire developed to assess a variety of dysfunctional beliefs thought to underlie OCD symptoms. Three factor analytically derived subscales correspond to the following domains of obsessive beliefs: (a) overestimates of threat and responsibility for harm, (b) importance and control of intrusive thoughts, and (c) perfectionism and the need for certainty. Participants rate their agreement with each of 44 statements from 1 (disagree very much) to 7 (agree very much). The instrument possesses good validity and internal consistency, and has been widely studied in clinical and nonclinical samples. Cronbach alphas for the subscales ranged from .89 to .91.
Session-level Change in Patient EX/RP Adherence Scale - Therapist Rated at each session beginning with session 4 | Sessions 4-16 (twice per week for 6 weeks following week 2 of treatment)
  The PEAS is a 3-item questionnaire that assesses patient adherence to between-session exposures and response prevention in exposure and response prevention (ERP) therapy. This form is rated by the therapist.
Treatment Credibility and Expectancy Questionnaire | Session 4 (2 weeks following Baseline)
  The Treatment Credibility and Expectancy Questionnaire is a 6-item questionnaire that assesses patient beliefs about the credibility and useful of the treatment they received, on a 10-point scale.
Change from Baseline Dimensional Obsessive Compulsive Scale (DOCS) at 8 weeks | Posttreatment (8 weeks after Baseline)
  The DOCS is a 20-item self-report measure that assesses the severity of the four most consistently replicated OCD symptom dimensions, which correspond to the measure's four empirically derived subscales: (a) contamination, (b) responsibility for harm and mistakes, (c) symmetry/ordering, and (d) unacceptable thoughts. Five items (rated 0 to 4) assess the following parameters of severity of each dimension: (a) time occupied by obsessions and rituals, (b) avoidance, (c) distress, (d) functional interference, and (e) difficulty disregarding the obsessions and refraining from rituals. Scores on these subscales converge well with other measures of OCD symptom dimensions. The internal consistency of the pre-treatment DOCS subscales in the present sample ranged from ( = .93-.96; total scale = .84).
Change from Posttreatment Dimensional Obsessive Compulsive Scale (DOCS) at 6 months | Follow-up (6 months after the end of treatment)
  The DOCS is a 20-item self-report measure that assesses the severity of the four most consistently replicated OCD symptom dimensions, which correspond to the measure's four empirically derived subscales: (a) contamination, (b) responsibility for harm and mistakes, (c) symmetry/ordering, and (d) unacceptable thoughts. Five items (rated 0 to 4) assess the following parameters of severity of each dimension: (a) time occupied by obsessions and rituals, (b) avoidance, (c) distress, (d) functional interference, and (e) difficulty disregarding the obsessions and refraining from rituals. Scores on these subscales converge well with other measures of OCD symptom dimensions. The internal consistency of the pre-treatment DOCS subscales in the present sample ranged from ( = .93-.96; total scale = .84).
Session-level Change in Dimensional Obsessive Compulsive Scale at each session | Sessions 1-16 (twice per week for 8 weeks following Baseline)
  The DOCS is a 20-item self-report measure that assesses the severity of the four most consistently replicated OCD symptom dimensions, which correspond to the measure's four empirically derived subscales: (a) contamination, (b) responsibility for harm and mistakes, (c) symmetry/ordering, and (d) unacceptable thoughts. Five items (rated 0 to 4) assess the following parameters of severity of each dimension: (a) time occupied by obsessions and rituals, (b) avoidance, (c) distress, (d) functional interference, and (e) difficulty disregarding the obsessions and refraining from rituals. Scores on these subscales converge well with other measures of OCD symptom dimensions. The internal consistency of the pre-treatment DOCS subscales in the present sample ranged from ( = .93-.96; total scale = .84).

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Twohig, Ph.D., Principal Investigator — Utah State University; Jonathan Abramowitz, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Utah State University, Logan, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data is available now.
Access Criteria: Data access requests should be directed to the one of the Principal Investigators via email. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Abramowitz JS, Deacon BJ, Olatunji BO, Wheaton MG, Berman NC, Losardo D, Timpano KR, McGrath PB, Riemann BC, Adams T, Bjorgvinsson T, Storch EA, Hale LR. Assessment of obsessive-compulsive symptom dimensions: development and evaluation of the Dimensional Obsessive-Compulsive Scale. Psychol Assess. 2010 Mar;22(1):180-98. doi: 10.1037/a0018260. PMID 20230164
- [Background] Abramowitz JS, Foa EB, Franklin ME. Exposure and ritual prevention for obsessive-compulsive disorder: effects of intensive versus twice-weekly sessions. J Consult Clin Psychol. 2003 Apr;71(2):394-8. doi: 10.1037/0022-006x.71.2.394. PMID 12699033
- [Background] Abramowitz JS, Franklin ME, Zoellner LA, DiBernardo CL. Treatment compliance and outcome in obsessive-compulsive disorder. Behav Modif. 2002 Sep;26(4):447-63. doi: 10.1177/0145445502026004001. PMID 12205821
- [Background] Abramowitz JS, Taylor S, McKay D. Potentials and limitations of cognitive treatments for obsessive-compulsive disorder. Cogn Behav Ther. 2005;34(3):140-7. doi: 10.1080/16506070510041202. PMID 16195053
- [Background] Abramowitz JS, Taylor S, McKay D. Obsessive-compulsive disorder. Lancet. 2009 Aug 8;374(9688):491-9. doi: 10.1016/S0140-6736(09)60240-3. PMID 19665647
- [Background] Beck, A. T. (1996). Beck Depression Inventory (2nd ed.). San Antonio, TX: The Psychological Corporation.
- [Background] Eifert, G. H., & Forsyth, J. P. (2005). Acceptance and commitment therapy for anxiety disorders: A practitioner's treatment guide to using mindfulness, acceptance, and values-based behavior change strategies. Oakland, CA US: New Harbinger Publications.
- [Background] Foa EB, Kozak MJ, Goodman WK, Hollander E, Jenike MA, Rasmussen SA. DSM-IV field trial: obsessive-compulsive disorder. Am J Psychiatry. 1995 Jan;152(1):90-6. doi: 10.1176/ajp.152.1.90. PMID 7802127
- [Background] Foa EB, Liebowitz MR, Kozak MJ, Davies S, Campeas R, Franklin ME, Huppert JD, Kjernisted K, Rowan V, Schmidt AB, Simpson HB, Tu X. Randomized, placebo-controlled trial of exposure and ritual prevention, clomipramine, and their combination in the treatment of obsessive-compulsive disorder. Am J Psychiatry. 2005 Jan;162(1):151-61. doi: 10.1176/appi.ajp.162.1.151. PMID 15625214
- [Background] Franklin, M. E. (2005). Combining serotonin medication with cognitive-behavior therapy: Is it necessary for all OCD patients. In J. Abramowitz & A. Houts (eds.). Concepts and controversies in obsessive-compulsive disorder (pp. 377-389). New York: Springer.
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Hayes, S. C. (2008). Climbing our hills: A beginning conversation on the comparison of acceptance and commitment therapy and traditional cognitive behavioral therapy. Clinical Psychology: Science and Practice, 15, 286-295.
- [Background] Hayes, S. C., Strosahl, K. D., & Wilson, K. G. (1999). Acceptance and commitment therapy: An experiential approach to behavior change. New York, NY US: Guilford Press.
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Kelley, M. L., Heffer, R. W., Gresham, F. M., & Elliott, S. N. (1989). Development of a modified Treatment Evaluation Inventory. Journal of Psychopathology and Behavioral Assessment, 11, 235-247.
- [Background] Leung AW, Heimberg RG. Homework compliance, perceptions of control, and outcome of cognitive-behavioral treatment of social phobia. Behav Res Ther. 1996 May-Jun;34(5-6):423-32. doi: 10.1016/0005-7967(96)00014-9. PMID 8687364
- [Background] Levitt, J. T., Brown, T. A., Orsillo, S. M., & Barlow, D. H. (2004). The effects of acceptance versus suppression of emotion on subjective and psychophysiological response to carbon dioxide challenge in patients with panic disorder. Behavior Therapy, 35, 747-766.
- [Background] Marcks BA, Woods DW. A comparison of thought suppression to an acceptance-based technique in the management of personal intrusive thoughts: a controlled evaluation. Behav Res Ther. 2005 Apr;43(4):433-45. doi: 10.1016/j.brat.2004.03.005. PMID 15701355
- [Background] Marcks BA, Woods DW. Role of thought-related beliefs and coping strategies in the escalation of intrusive thoughts: an analog to obsessive-compulsive disorder. Behav Res Ther. 2007 Nov;45(11):2640-51. doi: 10.1016/j.brat.2007.06.012. Epub 2007 Jul 5. PMID 17673167
- [Background] Masedo AI, Rosa Esteve M. Effects of suppression, acceptance and spontaneous coping on pain tolerance, pain intensity and distress. Behav Res Ther. 2007 Feb;45(2):199-209. doi: 10.1016/j.brat.2006.02.006. Epub 2006 Mar 29. PMID 16569396
- [Background] Paez-Blarrina M, Luciano C, Gutierrez-Martinez O, Valdivia S, Ortega J, Rodriguez-Valverde M. The role of values with personal examples in altering the functions of pain: comparison between acceptance-based and cognitive-control-based protocols. Behav Res Ther. 2008 Jan;46(1):84-97. doi: 10.1016/j.brat.2007.10.008. Epub 2007 Oct 22. PMID 18054894
- [Background] Simpson HB, Zuckoff AM, Maher MJ, Page JR, Franklin ME, Foa EB, Schmidt AB, Wang Y. Challenges using motivational interviewing as an adjunct to exposure therapy for obsessive-compulsive disorder. Behav Res Ther. 2010 Oct;48(10):941-8. doi: 10.1016/j.brat.2010.05.026. Epub 2010 Jun 1. PMID 20609435
- [Background] Steketee G, Chambless DL, Tran GQ, Worden H, Gillis MM. Behavioral avoidance test for obsessive compulsive disorder. Behav Res Ther. 1996 Jan;34(1):73-83. doi: 10.1016/0005-7967(95)00040-5. PMID 8561767
- [Background] Twohig MP, Hayes SC, Masuda A. Increasing willingness to experience obsessions: acceptance and commitment therapy as a treatment for obsessive-compulsive disorder. Behav Ther. 2006 Mar;37(1):3-13. doi: 10.1016/j.beth.2005.02.001. Epub 2006 Feb 21. PMID 16942956
- [Background] Twohig MP, Hayes SC, Plumb JC, Pruitt LD, Collins AB, Hazlett-Stevens H, Woidneck MR. A randomized clinical trial of acceptance and commitment therapy versus progressive relaxation training for obsessive-compulsive disorder. J Consult Clin Psychol. 2010 Oct;78(5):705-16. doi: 10.1037/a0020508. PMID 20873905
- [Background] Vogel, P. A., Stiles, T. C., & Gotestam, K. G. (2004). Adding cognitive therapy elements to exposure therapy for obsessive-compulsive disorder: a controlled study. Behavioural and Cognitive Psychotherapy, 32, 275-290.
- [Background] Woods, C. M., Chambless, D. L., & Steketee, G. (2002). Homework compliance and behavior therapy outcome for panic with agoraphobia and obsessive compulsive disorder. Cognitive Behaviour Therapy, 31, 88-95.